CLINICAL TRIAL: NCT06884124
Title: The Effect of Ventrogluteal Injection Training Using Microteaching Method on Students' Knowledge, Skills, and Anxiety Levels: a Randomized Controlled Trial
Brief Title: Effect of Microteaching on Ventrogluteal Injection Training
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ferhat Dasbilek, Teaching Assistant, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AU-SBF-FD-01
Record Dates: First submitted 2025-02-22; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Nursing Students; Intramuscular Injection
Keywords: nursing education; Micro-Teaching Method; Ventrogluteal Injection; Nursing Students

STUDY DESIGN:
Intervention Model Description: Title:
  Effect of Micro-Teaching Method on Knowledge, Skills, and Anxiety Levels in Ventrogluteal Injection Training for Nursing Students
  Study Design:
  This study is a randomized controlled trial designed to evaluate the effectiveness of the micro-teaching method on nursing students' knowledge, skills, and anxiety levels during ventrogluteal intramuscular (IM) injection training. The study will utilize a pre-test and post-test control group design to compare the outcomes between students receiving traditional teaching methods and those receiving micro-teaching intervention.
  Participants:
  The study will include undergraduate nursing students who are enrolled in the clinical practice course and have not previously received training in ventrogluteal IM injection.
  Intervention:
  The intervention group will receive ventrogluteal injection training using the micro-teaching method, which involves short, focused learning sessions enriched with interactive multimedia content and opportunities
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): In the control group, education will be conducted using routine lectures and a question-and-answer approach based on the learning objectives. Additionally, students in this group will observe the ventrogluteal injection procedure demonstrated on a mannequin in the laboratory setting, as per standard practice. After the demonstration, they will be asked to perform the procedure on the mannequin.
  Before the practice session, students will complete the "Ventrogluteal Injection Success Test and State Anxiety Inventory." After the practice, the "Ventrogluteal Injection Skill Evaluation Form" will be filled out by the instructor to assess the students' performance.
  In parallel with the intervention group, students in the control group will be asked to perform the procedure again one month later, and the "Ventrogluteal Injection Skill Evaluation Form" will be completed to evaluate their skill retention and improvement.
- Experimental (Experimental): During the first practice, students will be expected to prepare materials for the procedure, prepare medication according to the order, verify patient identity, identify the ventrogluteal injection site, and administer the medication at the ventrogluteal site. During the second practice, based on the feedback provided after the first session, students will be expected to improve themselves and their training by repeating the steps: preparing materials, preparing medication according to the order, verifying patient identity, identifying the ventrogluteal injection site, and administering the medication at the ventrogluteal site.
  Before the practice, students in the intervention group will be divided into subgroups. During the practice, each student in the subgroups will be expected to prepare for the following steps: material preparation, medication preparation according to the order, patient identity verification, identification of the ventrogluteal injection site, and administration
  Interventions: Behavioral: Experimental; Behavioral: Control

INTERVENTIONS:
Behavioral: Experimental — Micro teaching method will be applied for ventrogluteal injection training. Students will be trained with short learning units, multimedia content and feedback sessions.
  Arms: Experimental
Behavioral: Control — Routine lectures and practice will be done on the model
  Arms: Experimental

SUMMARY:
Nursing education plays a crucial role in ensuring nurses possess the necessary knowledge and skills to provide high-quality care. Inadequacies in knowledge and practical skills can compromise patient safety and negatively impact care quality. Therefore, integrating both theoretical and practical education that covers cognitive, psychomotor, and affective learning domains is essential for nursing students.

The micro-teaching method has emerged as an innovative educational approach, especially relevant for today's technology-savvy Generation Z students. It involves delivering small, focused learning units enriched with interactive multimedia content, which enhances knowledge retention, skill acquisition, and reduces student anxiety. This method also allows students to repeatedly access short videos and multimedia materials, enabling flexible and effective learning.

Intramuscular (IM) injection is a fundamental skill nursing students must master. Specifically, the ventrogluteal site is considered safer and more effective compared to the dorsogluteal site, as it is associated with fewer complications such as pain, bleeding, and nerve injury.

This study aims to examine the impact of ventrogluteal injection training using the micro-teaching method on nursing students' knowledge, skills, and anxiety levels. It is anticipated that this innovative educational approach will enhance learning outcomes, increase patient safety, and pave the way for future research in nursing education.

The study is unique as it explores an area that has not been previously investigated. Its findings are expected to contribute significantly to the literature, influencing the development of effective teaching methods not only in nursing education but also across other educational fields. Additionally, the study holds importance as it contributes to a doctoral thesis, highlighting its academic value.

DETAILED DESCRIPTION:
INTRODUCTION AND OBJECTIVE The educational processes of nurses are of great importance for the healthcare system; therefore, possessing the necessary knowledge and skills is essential for providing quality care (Atakoğlu et al., 2020). Deficiencies in knowledge and inadequacies in practical skills jeopardize patient safety and negatively impact the quality of care (Barisone et al., 2019). In this context, it is crucial to provide nursing students with both theoretical and practical training that integrates cognitive, psychomotor, and affective learning domains (Uysal, 2016; Tüzer et al., 2017; Yılmaz & Korhan, 2017).

Conducting nursing education both theoretically and practically is essential for students to effectively fulfill their roles in clinical settings and become competent professional nurses (Park et al., 2016). Reflecting theoretical knowledge into practice is also an integral part of students' education (Atakoğlu et al., 2020). It is emphasized that practical experiences facilitate knowledge retention, foster a deeper understanding, and enhance the permanence of learning (Rosencwaig, 2020). Therefore, nursing students should be provided with frequent practice opportunities to acquire the necessary psychomotor skills. These skills are typically taught in skills laboratories, where students have the opportunity to reinforce their theoretical knowledge through practice (Bayram & Çalışkan, 2019).

Students may also have the opportunity to practice in hospital clinics; however, this can bring about emotions such as fear of making mistakes, concern about harming patients, and feelings of inadequacy (Sezer & Orgun, 2017). Such experiences are among the most anxiety-inducing situations for students during clinical practice and education (Ross & Carney, 2017; Evgin et al., 2017).

With the expectations of today's technology-savvy Generation Z students and the advancements in information and technology in education, the use of innovative approaches and technology in nursing education has become essential (Güngör et al., 2023). Traditional theoretical lectures and laboratory demonstrations are insufficient to meet the needs of modern students (Stone et al., 2020). Therefore, educators are expected to develop innovative methods that facilitate students' retention of theoretical knowledge while ensuring patient safety (Butt et al., 2018).

Students' learning styles and needs have evolved with the integration of digital technologies into daily life (Carr et al., 2019). Microlearning has emerged as a teaching method that meets these new needs. Microlearning consists of small, focused learning units that are accessible through various devices (Lee, 2021). This method enriches lessons with interactive multimedia content and presents them in short durations. Students have the opportunity to access short videos and multimedia content repeatedly (Shail, 2019). These small learning components of microlearning allow students to decide what and when to learn, make connections between pieces of information, and enhance their knowledge and skills (Ahmad & Al-Khanjari, 2016; Anil & Slade Ogalo, 2012).

One of the essential skills nursing students need to acquire during their education is intramuscular (IM) injection application. Annually, over 12 billion medications are administered worldwide through IM injections (Vicdan et al., 2016). IM injections carry risks of complications such as chronic pain, necrosis, abscess, periostitis, and injuries to vessels, nerves, and bones (Kaya & Palloş, 2019; Lynn, 2015; Zaybak, 2023). Sciatic nerve injury is one of the most serious complications of IM injections, particularly resulting from injections in the dorsogluteal region (Kaya & Palloş, 2019). However, it has been reported that injections administered in the ventrogluteal region increase patient satisfaction and cause fewer complications such as bleeding, pain, and hematoma (İşseven, 2020; Apaydın & Öztürk, 2021).

In this context, it is crucial to equip nursing students with the skills to administer IM injections in the ventrogluteal region. Therefore, this study aims to determine the impact of ventrogluteal injection training provided through the micro-teaching method on nursing students' knowledge, skills, and anxiety levels.

ORIGINAL VALUE AND WIDESPREAD IMPACT This study will examine the effects of ventrogluteal injection training, delivered through the micro-teaching method, on nursing students' knowledge, skills, and anxiety levels. If the micro-teaching method is more widely adopted in educational processes, it could enhance educational effectiveness, benefiting nurses, individuals, and society.

The originality of this study is highlighted by the fact that this topic has not been addressed in previous research. The research aims to evaluate the effects of ventrogluteal injection training using micro-teaching on nursing students' knowledge, skills, and anxiety levels, thereby providing valuable data for future studies. The original values of the proposed study are as follows:

In terms of hypothesis: The proposed hypotheses are unique, as no previous studies have addressed this topic.

In terms of methodology: The study aims to determine the impact of ventrogluteal injection training using the micro-teaching method on students' knowledge, skills, and anxiety levels. No previous studies have been found that investigate the effects of such training on these parameters.

In terms of scientific quality: As the proposed project is original, it will contribute new knowledge to the literature.

The study plans to provide ventrogluteal injection training to students using the micro-teaching method, with the expectation that the findings will offer valuable insights for future research. If the study hypotheses are proven, the results will be easily applicable and cost-effective.

The absence of research comparing or applying the micro-teaching method in this context demonstrates the project's originality at both national and international levels. The findings will contribute to the literature by being published as scientific articles in high-impact journals and presented at national and international conferences, symposiums, and seminars. The knowledge gained from this project is expected to serve as a valuable resource not only for the nursing students in the study sample but also for other educational groups. Additionally, the study will pave the way for incorporating new methods into nursing education planning.

The originality and novelty of the research are expected to open the door to new studies and comparative research, thus contributing to the scientific literature. The advantages of different teaching methods will be observed, leading to the widespread use of innovative educational approaches. This will contribute to achieving the established standards in the quality of education provided to students. The findings from this project are expected to bring improvements to teaching methods and enhance the quality of nursing education.

The knowledge obtained from this project is anticipated to guide the selection of teaching methods, effectively enhancing the quality of nursing education. Improvements in students' interest and motivation, resulting in positive class participation, will be beneficial. The new knowledge gained from the project will lay the groundwork for future projects and contribute to the literature. Additionally, the widespread application of new methods across the country, as promoted by this project, could lead to significant advancements in education.

This study also holds importance as it constitutes a doctoral thesis.

ELIGIBILITY:
Inclusion Criteria:

* Graduated from Health Vocational High School,
* Have any previous experience with intramuscular injection,
* Repeating the "Nursing Principles" course,
* After graduating from the fields that provide associate degree education related to health, they are placed in the nursing department with the vertical transfer exam (DGS),
* No internet facility where they live,
* Students who do not want to participate in the study will be excluded from the study.

Exclusion Criteria:

* Incomplete responses to data collection forms,
* Who don't want to continue the research,
* Participants who are incomplete in at least one of the theoretical or practical phases of the study will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-06-02 (Estimated)

PRIMARY OUTCOMES:
Student Information Form | Pre-application
  This form was created by the researchers and consists of 7 questions to measure the demographic characteristics of the participants.
Ventrogluteal Injection Skill Evaluation Form | after the application, the student's video recording was monitored will be scored (Day 1 and 31)
  This form was prepared by the researcher based on the literature (Ay, 2015; Akbıyık, 2021, pp.535-551; Craven et al., 2015; Lynn, 2015; Süzen, 2015, pp.506-514) in order to evaluate the students' ability to administer IM injection to the ventrogluteal region and the form will be finalized by taking expert opinions. In the form, 33 procedures were listed for the steps of material preparation for the application, drug preparation in accordance with the order, patient identity verification, determination of the ventrogluteal injection site, and drug administration to the ventrogluteal injection site. For the content validity of the procedure steps, the opinions of 5 faculty members in the field of nursing principles and 3 faculty members who are experts in the field of teaching will be taken. The form will be applied to third year students because they have studied before. After the preliminary application of the form, item analysis will be performed for each question to determine the di
Ventrogluteal Injection Achievement Test | Before application
  This form was prepared by the researcher in line with the literature (Ay, 2015; Akbıyık, 2021, pp.535-551; Craven et al., 2015; Lynn, 2015; Süzen, 2015, pp.506-514) and the form will be finalized by taking expert opinions. The form contains an equal number of "True" and "False" statements. The form includes propositions that measure knowledge about ventrogluteal injection such as what ventrogluteal injection is, to which muscle it is applied, in which age group it can be applied, what to pay attention to before, during and after the injection. For the content validity of the questions, the opinions of 5 faculty members in the field of nursing principles and 3 faculty members who are experts in the field of teaching will be taken. The test will be administered to third year students because of their previous education. After the pre-application of the achievement test, item analysis will be performed for each question to determine the degree of difficulty and discrimination.
Micro Teaching Group Evaluation Form | will be used in the student's evaluation of the trainer after the training (Day 31)
  It was created by the researcher in line with the literature (Popovich & Katz, 2009; Göçer, 2016; Yang et al., 2019). The statements in the form consisting of 12 evaluations will be sent to the opinions of 3 instructors who are experts in the field of teaching. This form will be used both by the researcher and the peers in the same group to evaluate the training of the student practitioner.
State Anxiety Inventory | Before and one month after application
  This scale was first developed by Spielberg and colleagues (1970) and its validity and reliability study in Turkey was conducted by Öner and Le Compte (1983). The inventory consists of 20 items and asks individuals to describe how they feel at a certain time and under certain conditions, taking into account their feelings about their situation. In the scoring of the scale items, when the items indicating positive emotions are evaluated as "1" point, they are taken as "4" points, and when they are evaluated as "4" points, they are taken as "1" point. This scale was designed to measure the anxiety levels of individuals. In items related to positive emotions, a score of "1" symbolizes high anxiety and a score of "4" symbolizes low anxiety. On the other hand, for items involving negative emotions, a score of "4" indicates high anxiety, while low scores indicate a low level of anxiety. The 1st, 2nd, 5th, 8th, 10th, 10th, 11th, 15th, 16th, 19th, 19th and 20th items in the scale are reversib

CONTACTS AND LOCATIONS:
Overall Officials: Gülcin Avsar, Professor Doctor, Study Director — Ataturk University

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in this article, after de-identification (text, tables, figures, and appendices) will be shared. Data will be available beginning 6 months and ending 36 months following article publication to researchers who provide a methodologically sound proposal, to achieve the aims outlined in the approved proposal. Proposals should be directed to [your email].
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data and supporting information will be available 6 months after the publication of the study results and will be accessible for 3 years.
Access Criteria: Data will be available to researchers who provide a methodologically sound proposal that aims to achieve the objectives outlined in the approved research proposal. Access will be granted to researchers affiliated with academic institutions, research organizations, or healthcare organizations. Requests for data access should be directed to the principal investigator at [your email].